CLINICAL TRIAL: NCT05387044
Title: An Open-label, Phase II Single Arm Trial of SBRT for Oligoprogressive NSCLC After First Line Treatment With Immune Checkpoint Inhibitors
Brief Title: SBRT for Oligoprogressive NSCLC After First Line Treatment With Immune Checkpoint Inhibitors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Xiaojing Lai, Clinical Professor, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-OligoSBRT-IIT
Record Dates: First submitted 2022-05-13; First posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: NSCLC Stage IV
Keywords: NSCLC; Oligoprogressive; Immune checkpoint inhibitors; SBRT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT (Experimental): Patients with oligoprogressive NSCLC after first line treatment with immune checkpoint inhibitors will be treated with SBRT for all progressing lesions.
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — Patients with oligoprogressive NSCLC after first line treatment with immune checkpoint inhibitors will be treated with SBRT for all progressing lesions.

SUMMARY:
The treatment modality with immunotherapy has been the first-line standard treatment for advanced NSCLC. But more than 2/3 patients still develop acquired drug resistance within 5 years of immunotherapy, and more than 1/2 patients are oligoprogressive. Stereotactic body radiation therapy (SBRT) plays a growing role in the management of oligometastatic disease. This study aims to evaluate the efficacy and safety of SBRT for oligoprogressive NSCLC after first line treatment with immune checkpoint inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years;
* ECOG PS 0-1;
* Patients with pathologically confirmed stage IV NSCLC by tumor biopsy and/or fine-needle aspiration （AJCC the 8th Edition）;
* Stable Disease for at least 6 months after first line immunotherapy;
* Oligoprogressive disease in 5 or fewer lesions and 3 or fewer organs;
* All oligopreogressive lesion ≤ 5cm, and intracranial lesion ≤3cm or 30cc;
* Progressive disease would be amenable to SBRT and without indications for palliative radiotherapy in the opinion of the investigator;
* Patients with a history of radiotherapy are eligible if radiotherapy administered more than 4 weeks before study entry;
* Adequate organ function prior to enrollment:

Adequate bone marrow function: white blood cell (WBC) count ≥ 3.0 * 10 ^ 9/L or neutrophil count ≥ 1.5 * 10 ^ 9/L, platelet count ≥ 100 * 10 ^ 9/L and hemoglobin ≥90g/L,; Adequate hepatic function: total bilirubin, urea nitrogen and serum creatinine≤ 1.5 x upper limit of normal (ULN). Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤2.0 ULN;

* Life expectancy of more than 3 months;
* Ability to understand and willingness to provide the informed consent and signed informed consent for the use of fresh tumor biopsies before and during the treatment;
* Women of childbearing age and men must agree to use effective contraception during the trial.

Exclusion Criteria:

* History of another malignancy or concurrent malignancy (except for cured non-melanoma skin cancer, low-risk prostate cancer, T1/T2 glottic cancer, stage 0 or I breast cancer, non-invasive bladder cancer, cervical cancer in situ);
* Positive for driver genes including EGFR, ALK, and ROS-1;
* Mixed small cell with non-small cell lung cancer histology;
* Malignant pleural or ascites;
* Patients with brain metastasis require intracranial decompression;
* Symptoms of spinal cord compression;
* Severe autoimmune disease: inflammatory bowel disease (including Crohn's disease and ulcerative colitis), rheumatoid arthritis, scleroderma, systemic lupus erythematosus, Wegener's granulomatosis and related vasculitides;
* Symptomatic interstitial lung disease or clinically active infectious/non-infectious pneumonitis.
* History of another malignancy or concurrent malignancy;
* Active infection, congestive heart failure, or any evidence of myocardial infarction, unstable angina pectoris or cardiac arrhythmia within 6 months prior to enrollment;
* The patient is pregnant (confirmed by serum b-HCG if applicable) or is breastfeeding;
* Mental disorders, drug abuse, and social condition that may negatively impact compliance in the investigator's opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Progress free survival | two years
  PFS was defined from the date of enrollment to the date of disease progression

SECONDARY OUTCOMES:
Overall survival | two years
  OS was defined from the date of enrollment until death by any cause or last follow-up.
Grade 3 or higher toxicity | two years
  Treatment-related grade 3 or higher adverse events according to CTCAE 5.0.
Time to new metastasis | 2 years
  Time to new metastasis was defined from the date of enrollment to the date of new lesion progression.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojing Lai, Principal Investigator — Department of Thoracic Radiotherapy, Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No